CLINICAL TRIAL: NCT04467424
Title: TIVA With Ketofol Versus Lidoketofol for Short-term Anesthesia on Pediatric Patients; Effects on Recovery
Brief Title: Recovery After Total Intravenous Anesthesia With Ketofol Versus Mixture of Ketofol and Lidocaine for Short Pediatric Surgery
Acronym: Lidoketofol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Ana N Biliškov, MD, Pediatric anesthesiologist, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ketofol-Lidocaine
Record Dates: First submitted 2020-06-27; First posted 2020-07-13 (Actual); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Surgical Procedure, Unspecified
MeSH Terms: interventions — Ketamine; Propofol; Lidocaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pediatric anesthesia with ketofol (Experimental): ketamine, propofol
  Interventions: Drug: ketamine, propofol
- Pediatric anesthesia with ketofol plus lidocaine (Experimental): ketamine, propofol, lidocaine
  Interventions: Drug: ketamine, propofol, lidocaine

INTERVENTIONS:
Drug: ketamine, propofol — anesthesia with ketofol in pediatric surgery
  Arms: Pediatric anesthesia with ketofol
Drug: ketamine, propofol, lidocaine — anesthesia with ketofol plus lidocaine in pediatric surgery
  Arms: Pediatric anesthesia with ketofol plus lidocaine

SUMMARY:
Two hundred children aged 1-12 years undergoing short surgery will be randomized into two groups. Ketofol will be used for induction and maintenance of anesthesia in group l. .Ketofol with lidocaine will be prepared for group ll. A reducted McFarlan infusion dose will be used. Extubating time, duration of anesthesia, length of stay in post-anesthesia care unit (PACU) will be recorded.

DETAILED DESCRIPTION:
Aim of the research: In this study investigators want to examine the effectiveness of the use of ketofol and a mixture of ketofol and lidocaine on the total consumption of opioids and on the postoperative recovery of pediatric patients. Investigators will evaluate the safety, efficacy, and outcomes of the anesthesia procedure with respect to the administration of different anesthetics, specific pharmakocinetic profiles and compare the length of recovery between patients in two groups.

Including criteria: children aged 1 to 12 years who underwent short surgery (up to 60 min).

Primary and secondary outcome measures: The primary outcome of this study will be extubation time and the secondary outcome will be time spend in PACU.

Description of the study: Each subject included in the study will be given general anesthesia with ketofol or ketofol and lidocaine, with the addition of fentanyl. After 20 s the LMA will be placed. Maintenance of anesthesia will be performed using an air / oxygen mixture (50% / 50%) and an infusion of ketofol or ketofol and lidocaine. Ketofol will be prepare in a ratio of 1: 4 for induction and 1: 7 for maintenance. The same mixtures of ketofol will be added 1 ml of 2% lidocaine for the second group of patients. After extubation, patients will be transferred to the PACU.

ELIGIBILITY:
Inclusion Criteria:

* surgical procedures max 60 min ASA I and II

Exclusion Criteria:

* ASA > II surgical procedures longer than 60 min

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Split, Split, Croatia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pediatric Anesthesia With Ketofol | Pediatric Anesthesia With Ketofol Plus Lidocaine
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Age 1-12 years, male and female, for short surgery (max 60 min)
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric Anesthesia With Ketofol | Pediatric Anesthesia With Ketofol Plus Lidocaine | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants] — Age 1-12 years old, male and female, for short pediatric surgery (max 60 min.)
  Participants
    <=18 years | 100 | 100 | 200
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 78 | 81 | 159
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Croatia | 100 | 100 | 200
sevoflurane for iv cannula [Count of Participants; unit: Participants] | 64 | 54 | 118

OUTCOME MEASURES:

1. Primary Outcome: Effect of TIVA With Ketofol and Ketofol Plus Lidocaine on Extubation Time in Children
Time Frame: up to 600 seconds
Population: age 1-12, male and female, pediatric short surgery
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Pediatric Anesthesia With Ketofol | Pediatric Anesthesia With Ketofol Plus Lidocaine
Number analyzed (Participants) | 100 | 100
second | 240 [120 to 340] | 120 [41.5 to 170]

2. Primary Outcome: Effect of TIVA With Ketofol and Ketofol Plus Lidocaine on Length of Stay in the PACU
Time Frame: up to 40 minutes
Population: Age 1-12 years, male and female, pediatric short surgery
Measure: Median (Inter-Quartile Range); unit: minute
Arm/Group | Pediatric Anesthesia With Ketofol | Pediatric Anesthesia With Ketofol Plus Lidocaine
Number analyzed (Participants) | 100 | 100
minute | 35 [30 to 40] | 20 [20 to 25]

3. Secondary Outcome: Effect of TIVA With Ketofol and Ketofol Plus Lidocaine on Total Opioid Consumption
Time Frame: up to 60 minutes
Population: Age 1-12 years, male and female, pediatric short surgery
Measure: Median (Inter-Quartile Range); unit: microgram per kg
Arm/Group | Pediatric Anesthesia With Ketofol | Pediatric Anesthesia With Ketofol Plus Lidocaine
Number analyzed (Participants) | 100 | 100
microgram per kg | 2.3 [2 to 3] | 2.1 [2 to 2.8]

ADVERSE EVENTS:
Time Frame: 4 months
Description: NO adverse event.
Arm/Group | Pediatric Anesthesia With Ketofol | Pediatric Anesthesia With Ketofol Plus Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT04467424/Prot_SAP_000.pdf